CLINICAL TRIAL: NCT02041364
Title: Biomarkers of Fatigue Related to Adjuvant Chemotherapy for Breast Cancer: Evaluation of Plasma and Lymphocyte Expression.
Brief Title: Biomarkers of Fatigue Related to Adjuvant Chemotherapy for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, PhD, Faculdade de Medicina do ABC
Other Study IDs: Biomarker fatigue ABC001
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Fatigue; Breast Cancer
Keywords: Fatigue; Biomarkers; Breast Cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: patients without fatigue: Patients whose scores on the brief fatigue inventory (BFI) (15) won't increase after having received the first cycle of chemotherapy will be considered as controls
- Patients with fatighe: Patients whose scores on the brief fatigue inventory (BFI) (15) increase after having received the first cycle of chemotherapy will be considered as having manifested fatigue

SUMMARY:
Fatigue is common in cancer patients receiving adjuvant chemotherapy. To further understand the mechanism of fatigue and search for potential biomarkers, we will conduct a prospective study with breast cancer patients receiving adjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients with breast cancer undergoing adjuvant systemic chemotherapy based on the use of anthracyclines will be screened before the start of chemotherapy.

Patients whose scores on the brief fatigue inventory (BFI) increase after having received the first cycle of chemotherapy will be considered as having manifested fatigue. The patients whose fatigue won't worse following the first cycle of chemotherapy will be used as controls. We will collect blood samples of both groups before and 21 days after the start of chemotherapy. We will analyze the following biomarkers: IL2, IL10, TNF and TGFB-1 measured by amplification reaction; FSH, LH, estradiol, DHEA, DHEAS and cortisol hormones measured by chemiluminescent enzyme immunometric assay

ELIGIBILITY:
Inclusion Criteria:

* Non metastatic breast cancer;
* Patients undergoing adjuvant chemotherapy

Exclusion Criteria:

* hypothyroidism;
* Depression;
* anemia;
* heart disease or decompensated hypertension

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I, II and III breast cancer undergoing adjuvant systemic chemotherapy based on the use of anthracyclines will be screened before the start of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Potential biomarkers related to chemotherapy induced fatigue | 21 days after the start of chemotherapy
  This study examines potential biomarkers of fatigue induced by chemotherapy both in the plasma and mononuclear fraction of the peripheral blood of patients with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Felipe M Cruz, PhD, Principal Investigator — 551134744249
Locations (1):
- Cepho-Fmabc, Santo André, São Paulo, Brazil

REFERENCES:
- [Derived] Cruz FM, Munhoz BA, Alves BC, Gehrke FS, Fonseca FL, Kuniyoshi RK, Cubero D, Peppone LJ, Del Giglio A. Biomarkers of fatigue related to adjuvant chemotherapy for breast cancer: evaluation of plasma and lymphocyte expression. Clin Transl Med. 2015 Feb 14;4:4. doi: 10.1186/s40169-015-0051-8. eCollection 2015. PMID 25852820